CLINICAL TRIAL: NCT00382382
Title: Diffusion Tensor Imaging in Autism
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was completed but there were no participants. It was completed as a theoretical study. Requests for final progress report can be sent to Dr. Liu.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R03HD051656 (NIH)
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Autistic Disorder
Keywords: Autism; Asperger Syndrome; Restricted repetitive behavior; Stereotyped patterns of behavior; Typically Developing children; Human Volunteers
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Children with Autism (Other): A diffusion tensor imaging (DTI) will be done to examine the integrity of the white matter pathways in high functioning austistic children.
  Interventions: Other: diffusion tensor imaging (DTI)
- Healthy Volunteers (Other): A diffusion tensor imaging (DTI) will be done to examine the integrity of the white matter pathways in healthy volunteers.
  Interventions: Other: diffusion tensor imaging (DTI)

INTERVENTIONS:
Other: diffusion tensor imaging (DTI) — Both groups will have a diffusion tensor imaging (DTI) perform.

SUMMARY:
Using a new and more detailed approach to diffusion tensor imaging (DTI) recently developed in our lab, the investigators hope to learn more about irregularities in the brain that are related to autism. The investigators are especially interested in brain regions that contribute to repetitive behaviors in children with autism. Repetitive behaviors include stereotyped motor movements (hand-flapping), self-injurious behaviors (head hitting), compulsions (lining up toys), insistence on things staying the same, and difficulty with change. These behaviors often interfere with learning, can disrupt daily functioning, and can lead to other behavioral problems. Two specific aims will be accomplished:

Aim 1: To examine the integrity of white matter pathways in high functioning autistic children. The investigators hypothesize that autism is associated with specific white matter abnormalities in the cerebellum and other motor circuits. Additionally, the investigators expect to confirm and expand on previous reports of cerebral abnormalities by using newly developed DTI methods.

Aim 2: To determine whether there is a relationship between white matter abnormalities and the occurrence of restricted repetitive behaviors in children with autism. The investigators hypothesize that differences in the occurrence and type of restricted repetitive behaviors between autistic individuals are correlated with specific regional white matter abnormalities.

Results from the proposed experiments should contribute to current knowledge of brain abnormalities in autism and their relationship to restricted repetitive behaviors, and may be relevant to understanding the mechanisms underlying motor deficits in this disorder.

DETAILED DESCRIPTION:
Using a new and more detailed approach to diffusion tensor imaging (DTI) recently developed in our lab, the investigators aim to confirm and expand upon previous findings of white matter abnormalities throughout the brain in individuals with autism. The investigators have chosen to focus particularly on cerebellar and motor pathways in consideration of the prevalence of motor deficits in autism as well as brain structural studies that have indicated cerebellar abnormalities in autistic children. Finally, a proposal to investigate a possible functional association between white matter structure and the expression of restricted repetitive behaviors in autistic children, by correlating measures of white matter integrity with behavioral assessments indicating the severity of various forms of restricted repetitive behaviors. Two specific aims will be accomplished. Aim 1: To examine the integrity of white matter pathways in high functioning autistic children. The hypothesis is that autism is associated with specific white matter abnormalities in the cerebellum and other motor circuits. Additionally, it is expect to confirm and expand on previous reports of cerebral abnormalities by using newly developed DTI methods. Aim 2: To determine whether there is a relationship between white matter abnormalities and the occurrence of restricted repetitive behaviors in children with autism. The hypothesis is that differences in the occurrence and type of restricted repetitive behaviors between autistic individuals are correlated with specific regional white matter abnormalities. Results from the proposed experiments should contribute to current knowledge of brain abnormalities in autism and their relationship to restricted repetitive behaviors, and may be relevant to understanding the mechanisms underlying motor deficits in this disorder.

ELIGIBILITY:
Inclusion Criteria:

* male, aged 8-12 years of age
* clinical diagnoses of autism from a licensed professional for Autism or Asperger's Syndrome
* IQ >80
* no speech delay
* no major sensory or motor deficits

Exclusion Criteria:

* known genetic or medical conditions (e.g. Fragile X syndrome, tuberous sclerosis, Turner's syndrome)
* currently (within prior 3 months) taking anti-psychotic/dopamine-modulating medications

Ages: 8 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
RBS-R scores, including both total and subset scores | once

CONTACTS AND LOCATIONS:
Overall Officials: Mark H. Lewis, PhD, Study Director — University of Florida
Locations (1):
- McKnight Brain Institute of the University of Florida, Gainesville, Florida, United States